CLINICAL TRIAL: NCT02203994
Title: The Effect of Extracorporeal Shock Wave Therapy (ESWT) on Lower Limb Spasticity in Persons With an Incomplete Spinal Cord Injury
Brief Title: Extracorporeal Shock Wave Therapy (ESWT) for the Treatment of Spasticity in Persons With Spinal Cord Injury
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Cord Injury; Spasticity
Keywords: extracorporal shock wave therapy (ESWT); spasticity; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- extracorporeal shock wave therapy (ESWT) (Experimental): one-time treatment of the spastic muscle/ spastic muscles (adductor muscles and/ or M. triceps surae) with extracorporeal shock wave therapy (device: Duolith® SD 1 "T-Top" (Storz Medical AG, Tägerwilen, Switzerland))
  Interventions: Device: Duolith® SD 1 "T-Top" (Storz Medical AG, Switzerland)

INTERVENTIONS:
Device: Duolith® SD 1 "T-Top" (Storz Medical AG, Switzerland) — 2000 pulses per muscle, energy level: 0.030 mJ/mm2, frequency: 4 Hz

SUMMARY:
Spasticity is the most problematic self-reported secondary medical problem in patients with spinal cord injury. It has the potential to negatively influence quality of life through restricting activities of daily living. Problematic spasticity can cause pain and fatigue, disturb sleep, contribute to the developement of contractures and pressure ulcers, and has a negative effect on patients morbidity. For this reason there is enormous interest in therapeutic interventions addressing to decrease spasticity in persons with spinal cord injury. Recently, studies reported positive effects of extracorporeal shock wave therapy on spasticity in patients with stroke, focal limb dystonia and cerebral palsy. To date, no studies are published, assessing the effect of extracorporeal shock wave therapy on focal spasticity in patients with spinal cord injury.

The purpose of this study is to investigate the effect of a one-time ESWT on lower limb spasticity in patients with an incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non traumatic spinal cord injury
* Minimum age: 18 years
* Minimum time since spinal cord injury: two years
* Lesion: C3-Th10
* American Association of Spinal Cord Injury Impairment Score C and D
* Focal spasticity in the adductor muscles and/ or triceps surae
* Ability to walk 14 meters
* Spasticity/clonus/spasms disturbing the activities of daily living or participation

Exclusion Criteria:

* Changes in spasticity medication during the last 3 months
* Treatment with botulinum toxin during the last 6 months
* Anticoagulant medication
* Thrombosis
* Malignant tumors
* Pregnancy
* Inflammations or skin lesions in the treated area
* Acute urinary tract infection
* Intended change in spasticity medication within 5 days after intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
severity of spasticity | time 0, time 2h
  Ashworth Scale

SECONDARY OUTCOMES:
personal goal attainment | at day 0, 1, 3 and 5
  Goal Attainment Scale
walking speed | difference between pre- and post-intervention
  10 Meters Walking Test
walking distance | difference between pre- and post-intervention
  6 Minutes Walking Test
thickness of the treated muscle | difference between pre- and post-intervention
  thickness measurement of the treated muscle using ultrasound
severity of spasticity | time 0, time 2h
  Adductor Tone Rating Scale
severity of spasticity | time 0, time 2h
  Penn Spasm Frequency Scale
severity of spasticity | time 0, time 2h
  Clonus Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baumberger, Dr. med., Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland